CLINICAL TRIAL: NCT00622349
Title: A Phase III Randomised Study Comparing Three Combination Chemotherapy Regimens in Patients With Non Pre-treated Advanced Non-small Cell Lung Cancer
Brief Title: Randomised Study Comparing Three Chemotherapy Regimens in Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Lung Cancer Working Party (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ELCWP-01041
Record Dates: First submitted 2008-02-14; First posted 2008-02-25 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Randomised phase III; Chemotherapy; Advanced non-small cell lung carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Ifosfamide; Gemcitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental)
  Interventions: Drug: Cisplatin, Ifosfamide, Gemcitabine
- B (Active Comparator)
  Interventions: Drug: Ifosfamide, Gemcitabine
- C (Experimental)
  Interventions: Drug: Cisplatin, docetaxel

INTERVENTIONS:
Drug: Cisplatin, Ifosfamide, Gemcitabine — Cisplatin 50 mg/m² day 1 Ifosfamide 3g/m² day 1 (+ uromitexan rescue) Gemcitabine 1 g/m² days 1 and 8 Cycles every 3 weeks
  Arms: A
Drug: Ifosfamide, Gemcitabine — Ifosfamide 3g/m² day 1 (+ uromitexan rescue) Gemcitabine 1 g/m² days 1 and 8 Cycles every 3 weeks
  Arms: B
Drug: Cisplatin, docetaxel — Cisplatin 50 mg/m² day 1 Docetaxel 75 mg/m² day 1 Cycles every 3 weeks
  Arms: C

SUMMARY:
The purpose of this study is to determine if cisplatin-based chemotherapy, cisplatin-gemcitabine-ifosfamide or cisplatin-docetaxel, will improve survival in comparison to the combination gemcitabine-ifosfamide in patients with advanced NSCLC

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of non-small cell lung cancer
* Advanced (unresectable or functionally inoperable) stage III or stage IV disease
* Availability for participating in the detailed follow-up of the protocol
* Presence of an evaluable or measurable lesion
* Informed consent

Exclusion Criteria:

* Prior treatment with chemotherapy
* Operable patient with resectable tumour
* Performance status < 60 on the Karnofsky scale
* A history of prior malignant tumour, except non-melanoma skin cancer or in situ carcinoma of the cervix and cured malignant tumour (more than 5-year disease free interval)
* Polynuclear cells < 2,000/mm³
* Platelet cells < 100,000/mm³
* Serum bilirubin >1.5 mg/100 ml
* Serum creatinine > 1.5 mg/100 ml and/or creatinine clearance < 60 ml/min
* Perception hypoacousia
* Peripheral neuropathy
* Recent myocardial infarction (less than 3 months prior to date of diagnosis)
* Congestive cardiac failure requiring medical therapy or uncontrolled cardiac arrhythmia
* Uncontrolled infectious disease
* Serious medical or psychological factors which may prevent adherence to the treatment schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 707 (Actual)
Dates: Start 2004-02; Primary Completion 2009-03 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Survival | Survival will be dated from the first day of registration until death or last follow up

SECONDARY OUTCOMES:
Response rate | Every 3 courses of chemotherapy
Toxicity | After each course of chemotherapy
Activity of second-line chemotherapy | Every 3 courses of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Sculier, MD, PhD, Study Chair — European Lung Cancer Working Party
Locations (4):
- Department of Intensive Care Unit and Thoracic Oncology Institut Jules Bordet, Brussels, Belgium
- Pneumology department of CHU Lille, Lille, France
- Hellenic Cancer Institute - St Savas Oncology Hospital, Athens, Greece
- Medical Oncology Hospital de Sagunto, Valencia, Spain

REFERENCES:
- See also: Click here for more information on the protocol — http://www.elcwp.org
- See also: Trial registry of the French National Cancer Institute — http://www.e-cancer.fr